CLINICAL TRIAL: NCT03271840
Title: Registry for Primary Ciliary Dyskinesia: : Systematic Data Collection on Incidence, Clinical Presentation, Treatment and Course of the Disease
Brief Title: Registry for Primary Ciliary Dyskinesia
Status: Completed | Type: Observational
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: pro00074669
Record Dates: First submitted 2017-08-26; First posted 2017-09-05 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Primary Ciliary Dyskinesia
MeSH Terms: conditions — Ciliary Motility Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Primary Ciliary Dyskinesia (PCD) is a rare disease, which means that any single PCD center has experience with a limited number of patients. PCD Registry is the collection of data about PCD from many centers and countries who treat children with PCD. Collecting data about PCD increase the knowledge on PCD, better describe the course of the disease, and help to better understand the progression of the disease and be used to develop new treatments.

In the PCD registry of Alberta, important information about PCD such as time of diagnosis, symptoms, and tests which led to the diagnosis, state of health at diagnosis, the progression of lung function, the occurrence of severe infections, tests and treatments data will be collected from the patients' medical records.

DETAILED DESCRIPTION:
In order to better characterize the clinical course, and improve the diagnosis and treatment of PCD, the investigators propose to establish a provincial PCD registry in Alberta. This registry will be securely linked to the currently existing International Registry for PCD and will allow more researchers to use the information to do research on PCD.

The investigators will collect demographic data: current age, sex, age, diagnostic findings and symptoms at diagnosis; in addition, clinical data about PCD which are recorded during the past and future clinical visits and encounters (e.g. lung function, weight, height, infections, treatments, and complications) will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of PCD
* Abnormal findings in at least two of the following tests:

High-frequency video microscopic finding, transmission electron microscopy finding, immunofluorescence finding, low nasal NO concentration/production, demonstration of biallelic disease-causing mutations by genotyping.

Exclusion Criteria:

• Failure or unwillingness to give written informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with PCD
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2017-08-26 (Actual); Primary Completion 2021-11-25 (Actual); Study Completion 2021-11-25 (Actual)

PRIMARY OUTCOMES:
Age of diagnosis | 2017-2030
  Years
Lung Function | 2017-2030
  % predicted for age

CONTACTS AND LOCATIONS:
Overall Officials: Israel Amirav, MD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided